CLINICAL TRIAL: NCT00604240
Title: Telephone Follow-up From an Intensive Care Nursery: What do Parents Actually Remember?
Brief Title: Telephone Follow-up From an Intensive Care Nursery
Status: Completed | Type: Observational
Sponsor: Christiana Care Health Services (Other)
Collaborators: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Other Study IDs: 27164
Record Dates: First submitted 2008-01-17; First posted 2008-01-30 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Information Retention
Keywords: NICU; caregivers; discharge instructions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Parents / caregivers of any infant who has a length of stay of at least 1 week in the NICU at Christiana Hospital or Thomas Jefferson University Hospital.

SUMMARY:
The first few weeks after leaving the Neonatal Intensive Care Unit (NICU) can be a difficult transition time for caregivers of a previously hospitalized infant. To help ease this stressful period, doctors and nurses give caregivers a large amount of information prior to their infant leaving the NCIU. How much caregivers remember about medications, follow-up appointments, and general well-child care has not been studied. Caregivers who choose to participate will receive a phone call 2-7 days after discharge where they will be asked questions pertaining to the information that was discussed with them at the time of discharge. The purpose of the study is to determine how much information caregivers retain after leaving the NICU.

ELIGIBILITY:
Inclusion Criteria:

* Parents/caregivers of infants who have spent one week or longer in the NICU at Christiana Hospital or Thomas Jefferson University Hospital.

Exclusion Criteria:

* Parents / caregivers of infants who have spent less than one week in the NICU at Christiana Hospital or Thomas Jefferson University Hospital.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Parents/caregivers of infants who are hospitalized in the NICU
Sampling Method: Non-Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2007-11; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Amount of information that parents / caregivers are able to retain | Within one week after the infant is discharged from the NICU

CONTACTS AND LOCATIONS:
Overall Officials: Constance Andrejko, DO, Principal Investigator — Christiana Hospital and Thomas Jefferson University Hospital
Locations (2):
- United States (2):
  - Christiana Hospital, Newark, Delaware
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania